CLINICAL TRIAL: NCT05887362
Title: The Power of Hand Reflexology in Ameliorating Anxiety, Pain, and Fatigue Among Patients Undergoing Coronary Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Lecturer, Alexandria University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022935
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STUDY GROUP (Experimental): Each patient in the study group received 8 sessions of hand reflexology after CA in a room separating them from the patients in the control group.Using pleasant odourless almond oil to lubricate the patients' hands, the researcher used Ingham's approach to hand reflexology for 10 minutes, applying pressure for 5 minutes on the right hand and then the left.
  Interventions: Behavioral: Hand Reflexology
- Group 2 (No Intervention): The control group was selected first and received the routine care delivered by the hospital, such as assessment of vital signs, supine position, complete bed rest, and hygienic care. They didn't receive the hand reflexology intervention.

INTERVENTIONS:
Behavioral: Hand Reflexology — Reflexology is a well-known, safe, and noninvasive alternative medicine technique. It alludes to a treatment that is applied to particular areas of the hands and feet. The compression on the hands or feet serves as a sensor linked to particular body areas. These sensors are activated by the reflexology technique to improve blood flow, energize, relax, and maintain homeostasis.
  Arms: STUDY GROUP

SUMMARY:
Reflexology influences pain perception and pain-impulse transmission by releasing endorphins (12). Patients with a variety of medical illnesses can benefit from hand reflexology by lessening their physical and emotional discomfort (13, 14). Therefore, this study was done to investigate the power of hand reflexology in ameliorating anxiety, pain, and fatigue among patients undergoing coronary angiography

ELIGIBILITY:
Criteria:

Inclusion Criteria:

* Patients between the ages of 20 and 60 who were scheduled for non-emergency CA, Absence of any hands' sensory motor disorders, or upper limb vascular injuries.
* No abnormalities such as amputations, burns, skin lesions, and intervertebral disc herniation.
* No history of mental illnesses.

Exclusion Criteria:

Patients with severe mental problems

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 4 months
  It is a 10 cm horizontal line with two ends; the left end typically denotes "no pain," while the right end typically denotes "worst possible pain."
Fatigue | 4 months
  The Rhoten Fatigue Scale (RFS) is a subjective rating scale developed by (16) to measure a patient's fatigue level. It comprises a 10-centimeter line with extremely positive and negative statements at either end.
Anxiety | 4 months
  The Beck Anxiety Inventory (BAI) was developed in 1988 by (17) to assess the severity of anxiety symptoms. The Likert scale for the 21 items that comprise the BAI ranges from 0 to 3. The overall score is between 0 and 63.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ali EA, Awad WHA, Khedr MA, Rabie EAEGA. Effect of hand reflexology in ameliorating anxiety, pain, and fatigue among patients undergoing coronary angiography. BMC Complement Med Ther. 2023 Nov 24;23(1):425. doi: 10.1186/s12906-023-04256-6. PMID 38001461